CLINICAL TRIAL: NCT01381783
Title: Phacoemulsification Under Topical Anesthesia and Its Complications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Oftalmologia Ivo Correa-Meyer (Other)
Responsible Party: Manuel Augusto Pereira Vilela, Instituto de Oftalmologia Ivo Correa-Meyer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: facectopica
Record Dates: First submitted 2011-04-07; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-03

CONDITIONS: Phacoemulsification
Keywords: topical anaesthesia; Phacoemulsification
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical anesthesia (Other)
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Procedure: Phacoemulsification — Phacoemulsification under topical anesthesia

SUMMARY:
The purpose of this study is to determine if topical anesthesia is safe for phacoemulsification in eyes with comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* patients with cataract with a visual acuity less than 0.8

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Number of Postoperative events | 12 months
  To describe any postoperatives events in a phacoemulsification surgery under topical anesthesia